CLINICAL TRIAL: NCT05813509
Title: Chief Physician of Obstetrics and Gynecology Department of the First Affiliated Hospital of Xiamen University
Brief Title: Individualized Precision Treatment Based on Ovarian Cancer Organoid Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMYY-2022KY110
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2022-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer；Platinum-resistant；chemosensitivity
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Platinum resistant ovarian cancer (Experimental): Advanced-stage epithelial ovarian cancer (stage III or above) that has received more than 2 lines of chemotherapy and recurred within 6 months after the chemotherapy is stopped;
  Interventions: Device: Organoid culture

INTERVENTIONS:
Device: Organoid culture — Tumor like organ is a kind of organ cultured from tissues of tumor patients, which is a small tumor growing in a culture dish. Compared with the traditional two-dimensional culture system, the most important feature of this technological innovation is that it can directly use the patient's own tissue to culture organ like cells. At the same time, these organ like cells can well replicate some key characteristics of the primary tumor and retain the pathological form and biological mechanism of the patient's tissue

SUMMARY:
The research purpose of this study is to use organoid cultured from patients' own ovarian cancer tissues as models, screen potential clinical therapeutic drugs (such as paclitaxel, gemcitabine, etc.) in vitro, formulate individualized drug treatment plans for individual patient, and evaluate the clinical application value of organ like drug sensitivity technology.

DETAILED DESCRIPTION:
Under the guidance of ultrasound, the lesions were punctured to obtain tumor cells; The cells were amplified and cultured by organ like culture method to establish ovarian cancer like organoid. The drug sensitivity tests of different drugs were carried out on similar organs. Number of drugs tested: 10 (paclitaxel, carboplatin, lobaplatin, doxorubicin, etc.); After the test is completed, sufficient chemotherapy for full course of treatment shall be carried out according to the drug sensitivity results; After chemotherapy, blood and imaging evaluation were performed; Collect the information of patients from initial treatment to the end of chemotherapy; Matching the corresponding number of patients with platinum resistant relapse who did not undergo organ like culture; At each end point, the evaluation and comparison were carried out and the research conclusions were drawn.

ELIGIBILITY:
Inclusion criteria

1. Patients diagnosed as primary nonmucous epithelial ovarian cancer with stage III or above by previous pathological diagnosis;
2. According to the relevant standards formulated by the World Health Organization (WHO) in 2014, measurable or assessable lesions are determined;
3. platinum-resistant epithelial ovarian cancer that has received more than 2 lines of chemotherapy;
4. There is no serious disease of important organs, and the patient can tolerate chemotherapy. Karnofsky score more than 60, and the expected survival period is more than half a year;
5. The liver, kidney and bone marrow functions were good.

Exclusion criteria

1. Patients with other malignant tumors;
2. Patients with nervous system diseases;
3. Hepatitis B virus and human papilloma virus infection;
4. Immune function defect or serious infection;
5. Patients who cannot communicate effectively, disagree with the research requirements, and do not understand the research purpose.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate | 6 months
  partial or complete remission ratio according to RECIST criteria

SECONDARY OUTCOMES:
Progression free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China